CLINICAL TRIAL: NCT05852015
Title: Digital Mindfulness-Based Treatment for Individuals in Early Recovery From Substance Use Disorders
Brief Title: Digital Mindfulness-Based Treatment for Substance Use Disorder Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Corey Roos, Assistant Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000028537; 1K23AT011342-01 (NIH)
Record Dates: First submitted 2023-04-17; First posted 2023-05-10 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment-as-Usual (TAU) (Active Comparator): TAU consists of weekly outpatient-based group therapy
  Interventions: Behavioral: Treatment-as-Usual (TAU)
- TAU Plus Digital Mindfulness-Based Treatment (Experimental): TAU consists of weekly outpatient-based group therapy. The digital mindfulness-based treatment is multimedia app-based program teaching mindfulness skills.
  Interventions: Behavioral: Treatment-as-Usual (TAU); Behavioral: Digital Mindfulness Treatment

INTERVENTIONS:
Behavioral: Treatment-as-Usual (TAU) — TAU consists of weekly outpatient-based group therapy for substance use disorder
Behavioral: Digital Mindfulness Treatment — The digital mindfulness-based treatment is a multimedia app-based program teaching mindfulness skills to facilitate recovery from substance use disorder
  Arms: TAU Plus Digital Mindfulness-Based Treatment

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility and acceptability of a digital mindfulness-based treatment for individuals in early recovery from substance use disorders. Participants are randomized to treatment-as-usual (TAU) or TAU plus the digital mindfulness-based treatment. The digital treatment will be completed over an 8-week period.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Fluent in English and have a 6th grade or higher reading level
* Have completed 1 month or more of SUD treatment
* Report use of their primary substance of choice in past 6 months
* Are not currently enrolled in residential/inpatient treatment
* Are willing to be randomized
* Are willing and able to participate for the entire study period
* Are willing to provide locator information for follow-up
* Own a working, WIFI-enabled smartphone

Exclusion Criteria:

* Current psychotic disorder
* High suicide risk characterized by suicidal ideation with intent
* Homicidal ideation posing imminent danger to others
* Pending legal case, imminent incarceration, or a planned move that results in inability to commit to procedures during the entire study period
* Participation in the Phase 1 User Testing study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Adherence to the digital treatment | 8-week treatment period that begins on the day participants are randomized
  Percent of randomized participants completing 50% or more of the digital treatment modules
Completion rates for the post-treatment assessment visit | Approximately 9 weeks after randomization
  Percent of randomized participants completing post-treatment assessment visit
Completion rates for the follow-up assessment visit | 2-month post-treatment follow-up (approximately 16 weeks post-randomization)
  Percent of randomized participants completing follow-up assessment visit
Completion rates for ecological momentary assessment at baseline | 2-week period at baseline prior to randomization
  Percent of randomized participants completing 50% or more of EMA surveys at baseline
Completion rates for ecological momentary assessment at post-treatment | 2-week period occurring approximately during weeks 10 and 11 post-randomization
  Percent of randomized participants completing 50% or more of EMA surveys post-treatment
Dimensions of treatment acceptability | Ratings made at the post-treatment assessment, which is approximately 9 weeks after randomization
  Single-items measuring ratings of acceptability dimensions for the digital treatment, including willingness to engage, usability, understandability, engage-ability, visual appeal, helpfulness, skill acquisition, and confidence implementing skills. Scores for each item range from 1 to 5, with higher scores indicating better acceptability.

OTHER OUTCOMES:
Change in frequency of primary substance use | Baseline through end-of-treatment (end of week 8 post-randomization) and through the 2-month follow-up period (weeks 9 to 16 weeks post-randomization)
  The Timeline Follow Back, a calendar-based interview, will be used to assess substance use
Change in frequency of any substance use | Baseline through end-of-treatment (end of week 8 post-randomization) and through the 2-month follow-up period (weeks 9 to 16 weeks post-randomization)
  The Timeline Follow Back, a calendar-based interview, will be used to assess substance use
Change in substance-related problems | Baseline through end-of-treatment (end of week 8 post-randomization) and through the 2-month follow-up period (weeks 9 to 16 weeks post-randomization)
  Short-inventory of problems Revised (SIP-R), a self-report questionnaire of substance-related problems. Total score range from 0 to 51, with higher scores indicating greater substance related problems.

CONTACTS AND LOCATIONS:
Locations (1):
- 1 Church street, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests for data sharing will be considered within the context of ongoing and planned research being performed within the research group at Yale in order to avoid duplication of effort and overlap in data analysis that might compromise communication of findings. Data to be shared will be de-identified and transmission electronically and securely, as we have done previously with investigators at other institutions.